CLINICAL TRIAL: NCT01660503
Title: Dose Response Effects of Soluble Corn Fiber (SCF) on Calcium Metabolism and Gastrointestinal Microflora in Adolescents
Brief Title: Dose Effects of SCF on Calcium Metabolism and GI Microflora in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Tate and Lyle Ingredients Americas LLC (Unknown)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Tate & Lyle Teen Study
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
Keywords: Calcium absorption; Osteoporosis; Bone Health; Adolescent
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- No SCF (Placebo Comparator): Twice daily consumption of snack foods containing no SCF.
  Interventions: Dietary Supplement: 0 grams SCF
- 10 grams SCF (Experimental): Twice daily consumption of snack foods, each containing 5 grams SCF
  Interventions: Dietary Supplement: 10 grams SCF
- 20 grams SCF (Experimental): Twice daily consumption of snack foods, each containing 10 grams SCF
  Interventions: Dietary Supplement: 20 grams SCF

INTERVENTIONS:
Dietary Supplement: 0 grams SCF — Given in snack foods (muffins and flavored beverage)
  Arms: No SCF
Dietary Supplement: 10 grams SCF — Given in snack foods (muffins and flavored beverage)
  Arms: 10 grams SCF
Dietary Supplement: 20 grams SCF — Given in snack foods (muffins and flavored beverage)
  Arms: 20 grams SCF

SUMMARY:
Soluble corn fiber (SCF) has been shown to enhance calcium utilization and bone properties in rats and in adolescent boys and girls.

DETAILED DESCRIPTION:
The growing knowledge of non-digestible oligosaccharide (NDO)-related health benefits has led to the identification of other fermentable carbohydrates which may improve bone balance and bone health parameters. One such carbohydrate is the corn derivative, soluble corn fiber (SCF). Already known for its association with improved intestinal health and influence on colonic microflora content, we have been studying the effects of SCF on calcium absorption and bone health. First we found that soluble corn fiber (SCF) greatly enhanced calcium utilization and bone properties in a growing rat model. Results from this study demonstrated that SCF was capable of increasing bone mineral content, density and bone strength parameters in 4-week old, male rats. Our study in adolescent boys and girls showed a 12% increase in calcium absorption after consuming 12 g SCF for 21 days compared to a control period in a crossover design using a controlled feeding metabolic balance approach. Given these profound changes on calcium absorption and in bone, a logical next step is to study a dose-response effect of SCF on calcium absorption, bone turnover, and gut microflora in free-living adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescent Caucasian girls between the ages of 12-14. This population has been chosen because they exhibit higher risk for osteoporosis later in life.

Exclusion Criteria:

* Habitual dietary patterns including less than 550 and greater than 1500 mg Ca per day. This represents the 5th and 95th percentile of usual intake of girls 9-13 y in the US.
* History of smoking, alcohol use, illegal or non-prescription drug use
* History of disordered calcium or bone metabolism e.g. Paget's disease, hyper or hypo-calcemia
* History of gastrointestinal diseases (Crohn's, celiac, inflammatory bowel disease)
* History of diseases that affect kidney or liver function.
* Body Mass Index (BMI) less than 5th percentile for age or greater than the 90th percentile for age
* Having a broken bone within the last 6 months.
* Regular consumption of foods or supplements containing prebiotics or probiotics
* History of pregnancy or use of contraceptives

Ages: 9 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Calcium Absorption | 4 Weeks
  The subject will be asked to consume one snack item in the morning and one snack in the evening for four consecutive weeks.
  After consuming the SCF product for four weeks the teen will come to Purdue University campus for 3 nights and days (e.g. Thursday noon - Sunday noon). They will reside in university residence hall or hotel near campus. Calcium Absorption testing will be done utilizing 43Ca and 44Ca.

SECONDARY OUTCOMES:
GI microbial changes | 4 weeks
  Fecal microbial analyses will be performed on a baseline sample collected before each 4 week consumption period to establish basal microbial profiles. Additional analyses will be performed on fecal samples collected during the 3 day clinical visit to compare microbial changes in response to SCF treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, Ph.D., Principal Investigator — Purdue University; Berdine R Martin, PhD, Study Director — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Whisner CM, Martin BR, Nakatsu CH, Story JA, MacDonald-Clarke CJ, McCabe LD, McCabe GP, Weaver CM. Soluble Corn Fiber Increases Calcium Absorption Associated with Shifts in the Gut Microbiome: A Randomized Dose-Response Trial in Free-Living Pubertal Females. J Nutr. 2016 Jul;146(7):1298-306. doi: 10.3945/jn.115.227256. Epub 2016 Jun 8. PMID 27281813